CLINICAL TRIAL: NCT04665596
Title: Prospective, Controlled, Single-arm Clinical Investigation for the Treatment of Subjects With Severe Symptomatic Aortic Valve Stenosis Using Valvosoft® Pulsed Cavitational Ultrasound Therapy (PCUT) - First-In-Human
Brief Title: Valvosoft First-In-Human Study in Severe Symptomatic Aortic Stenosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiawave SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CW19-01RS
Record Dates: First submitted 2020-11-23; First posted 2020-12-11 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Aortic Valve Stenosis
Keywords: symptomatic; aortic valve; stenosis; ultrasound; non-invasive
MeSH Terms: conditions — Aortic Valve Stenosis; Constriction, Pathologic

STUDY DESIGN:
Intervention Model Description: Ultrasound treatment of calcific aortic stenosis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound treatment (Experimental): Ultrasound treatment of patients with symptomatic aortic valve stenosis who are not eligible for valve replacement
  Interventions: Device: Ultrasound treatment

INTERVENTIONS:
Device: Ultrasound treatment — Ultrasound treatment of calcified aortic valve causing symptomatic aortic valve stenosis in patients who are not eligible for valve replacemen
  Other Names: Ultrasound treatment of calcific aortic valve

SUMMARY:
This is a prospective, controlled, single-arm clinical investigation for the treatment of subjects with severe symptomatic aortic valve stenosis using Valvosoft® Pulsed Cavitational Ultrasound Therapy (PCUT) - First-In-Human

DETAILED DESCRIPTION:
CARDIAWAVE has developed a new non-invasive, real-time image-guided, therapeutic approach to treat patients suffering from Calcified Aortic Stenosis. CARDIAWAVE's Valvosoft device is a new ultrasound therapy based on a disruptive technology involving delivering an extremely precise and focused ultrasound beam to perform a reparative effect on the aortic valve leaflets, softening the valve's tissues, restoring leaflet mobility, and therefore improving the overall clinical status related to the aortic valve stenosis. In this study, a brai-MRI is performed before the procedure and 24-72 hours after the procedure to detect cerebrovascular events.This is a FIM study

ELIGIBILITY:
Inclusion Criteria:

* Subjects suffering from severe symptomatic aortic valve stenosis according to ESC 2017 definition, including subjects with a bicuspid valve.
* Patient is not eligible for TAVR/SAVR according to local Heart Team.
* Age ≥18 years.
* Subjects who are willing to provide a written informed consent prior to participating in the study.
* Subjects who can comply with the study follow up or other study requirements.
* Patient is eligible for the Valvosoft procedure according to CRC.

Exclusion Criteria:

* Subjects with any electrical device implanted.
* Subjects with unstable arrhythmia not controlled by medical treatment.
* Subjects with implanted mechanical valve in any position or bio prosthetic valve in aortic position.
* Subjects with complex congenital heart disease.
* Chest deformity.
* Cardiogenic shock.
* History of heart transplant.
* Subjects requiring other cardiac surgery procedures (bypass graft surgery, mitral valve procedure, tricuspid valve procedure) within one month after treatment.
* Thrombus in heart.
* Acute myocardial infarction (MI), stroke or transient ischemic attack (TIA) within one month prior to enrolment*.
* Subjects who are pregnant or nursing.
* Subjects who are participating in another research study for which the primary endpoint has not been reached.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Safety: Rate of procedure related mortality | Up to 30 days
  Rate of procedure related mortality at 30 days
Device performance to modify valve structure as measured by echocardiography | Immediately after the procedure
  Ability to modify the Left Ventricular Ejection Fraction (%)
Device performance to modify valve structure as measured by echocardiography | Immediately after the procedure
  Ability to modify the Mean Pressure Gradient (mmHg)

SECONDARY OUTCOMES:
All-cause mortality | Up to two years
  Number of patients that die during the course of the study and if so, how long aftre the procedure
Rate of stroke | Up to two years
  Rate of stroke
Change of severity of heart failure | At 1, 3,6,12 and 24 months
  Change of New York Heart Association class (I-IV - stage of severity of heart failure - I=no symptoms, IV= symptoms at rest)
Major Adverse Events | Up to 2 years
  Rate of Major Adverse Events (MAE) and number of patients with one or more MAE during the course of the study, an MAE defined as: Disabling stroke, Myocardial infarction or any clinically significant changes in biomarkers (CK, Troponin I - T) that would indicate damage to the heart structure, or clinically significant conduction disturbances requiring pacemaker implantation or persistent arrhythmias
Adverse events | Up to 2 years
  Rate of all Adverse Events
User Handeling | Immediately after the procedure
  User handling (questionnaire for operator + procedure duration
Long term maintenance of improvement of Aortic Valve area and mean Pressure Gradient | At 1, 3, 6,1 2 and 24 months
  Long term maintenance of improvement of AVA and PG
quality of life measured through Kansas City Cardiomyopathy Questionnaire | at 1, 3, 6, 12 and 24 months
  Improvement of quality of life by means of KCCQ

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel Messas, MD, Principal Investigator — Hospital Georges Pompidou, Paris, France
Locations (1):
- Clinical Centre of Serbia, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trifunovic-Zamaklar D, Velinovic M, Kovacevic-Kostic N, Messas E. Systematic brain magnetic resonance imaging and safety evaluation of non-invasive ultrasound therapy for patients with severe symptomatic aortic valve stenosis. Eur Heart J Cardiovasc Imaging. 2023 Jun 21;24(7):e108-e109. doi: 10.1093/ehjci/jead089. No abstract available. PMID 37158997
- [Background] Messas E, Ijsselmuiden A, Trifunovic-Zamaklar D, Cholley B, Puymirat E, Halim J, Karan R, van Gameren M, Terzic D, Milicevic V, Tanter M, Pernot M, Goudot G. Treatment of severe symptomatic aortic valve stenosis using non-invasive ultrasound therapy: a cohort study. Lancet. 2023 Dec 16;402(10419):2317-2325. doi: 10.1016/S0140-6736(23)01518-0. Epub 2023 Nov 14. PMID 37972628